CLINICAL TRIAL: NCT03523923
Title: The Effectiveness of Collaborative Care Versus Usual Care for Pain After Traumatic Brain Injury
Brief Title: TBI Care: Collaborative Care for Pain After Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor, School of Medicine: Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003847
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Brain Injuries, Traumatic; Chronic Pain; Post-Traumatic Headache
Keywords: Collaborative Care; Effectiveness Study
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Pain; Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: Randomized, 1:1 controlled trial effectiveness study comparing Collaborative Care (CC) to usual care (UC) to reduce pain interference among outpatients in our UW Medicine TBI clinics who have chronic pain, including headache, and meet other eligibility criteria.
Who Masked: Outcomes Assessor
Masking Description: This study uses masked outcome assessments; research staff members who collect outcome data from participants at 4 and 8 months must be unaware of participants' treatment group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): If assigned to the Usual Care (UC) arm, participants receive the same care as they would normally received from the HMC or UWMC outpatient TBI clinics, which could include similar types of treatment (medication changes, referral to specialists, etc.).
- Collaborative Care (Active Comparator): If assigned to the Collaborative Care (CC) arm, participants receive up to 12 sessions (45-60 minutes) of scheduled contacts with a Collaborative Care Manager (CCM) over 16 weeks of treatment. The CCM meets weekly for supervision with a team of experts to determine appropriate care.
  Interventions: Behavioral: Collaborative Care

INTERVENTIONS:
Behavioral: Collaborative Care — Up to 12 phone sessions over 16 weeks from Collaborative Care Manager (CCM).
  Session 1: Establish rapport, perform structured clinical assessment explain the rationale and parameters of the intervention, provide brief education on pain and together with the participant create an overall treatment plan and detailed follow-up plan.
  Sessions 2-12 Components:
  * Care Management Weekly monitoring of response to treatment using standardized measures.
  * Collaborative Medical Management: Optimized management of problem areas. Medication recommendations will follow evidence-based treatment algorithms with consultation of supervisors.
  * Psychosocial Treatment: Evidence based, focus on pain self-management skills/education, initially on foundational skills including: (1) pain education; (2) relaxation skills training; (3) behavioral activation and goal setting; 4) importance of physical activity and (5) motivational interviewing to promote adherence to healthcare and goals.
  Arms: Collaborative Care

SUMMARY:
The purpose of this study is to (1) test the benefits of the patient-centered collaborative care treatment approach for persons who have had a TBI and who have pain, including headache; and also (2) test whether this approach improves quality of life, patient satisfaction, adherence to other treatments, and quality of care in the TBI care system.

This project uses the contextual paradigm of disability to analyze and improve outpatient treatment of pain, including headache, in people who have had a TBI. Issues of restricted access and health care system complexity likely contribute to sub-optimal treatment of chronic pain. Therefore, the investigators seek to enhance real-world outpatient healthcare delivery through a patient-centered, collaborative care approach to treating chronic pain. The intervention is structured to reduce pain interference directly and indirectly through improved management of pain and comorbid conditions (e.g., depression, anxiety, and sleep difficulties) that can amplify pain perception and disability. In addition, change in the system of care may reduce burden on the emergency department. The investigators have heard from our clinician and patient partners that poor pain management often leads to emergency department visits, and this has also been reported in the literature.

DETAILED DESCRIPTION:
Screening

Potential participants may be referred to the study by clinical staff, self-refer based on seeing study brochures or flyers, or will be invited to participate based on review of medical records of patients scheduled for TBI clinics at Harborview Medical Center (HMC) or the University of Washington Medical Center (UWMC) Rehabilitation TBI clinics.

If a potential participant meets initial eligibility criteria of having a diagnosis of TBI and reports of chronic pain, a research staff member will contact the patient to confirm eligibility through a formalized Institutional Review Board (IRB)-approved screening questionnaire. The Six-Item Screener (a brief and reliable instrument for identifying cognitive impairment) will be used to determine if the participant is cognitively able to provide informed consent.

Once eligibility is confirmed, research staff will introduce the study using a talking points script, and if the potential participant is interested, provide a brochure and a consent form. Potential participants will be fully informed of all risks and benefits prior to giving their written informed consent and prior to enrollment in the study. They may take time to think about participating and render a decision in a subsequent call or visit. Potential participants will be asked to repeat back understanding of this material as necessary.

Research staff will also review a HIPAA authorization form with the participant that permits research staff to collect data from the participant's medical records regarding injury and medical history.

The investigators plan to enroll a total of 158 participants with the goal of outcomes assessment on 63 subjects in each arm (total of 126).

Basic Demographic Information

Basic demographic information including age, sex, and race will be collected via medical record review without consent from all patients including those who do not enroll to determine differences between enrolled patients participants and those who do not enroll to examine potential bias.

Procedures

Randomization

Once enrolled, participants will be randomized into one of two groups: usual care (UC) or Collaborative Care (CC). Those randomized to CC treatment group will work with Collaborative Care Manager (CCM) for up to 12 contacts over a 16 week treatment period, and complete a 24 week post randomization check in call with CCM.

Participants assigned to the UC arm will be informed of the assignment via phone by an un-blinded research team member. In addition, participants assigned to the UC arm will receive a letter explaining the assignment. Participants assigned to the CC arm will be contacted by the CCM to arrange the timing of their first treatment session.

Data Collection

Participants may choose to have the interview/s administered by phone or in person at either UWMC or HMC by our research staff member.

Baseline Interview:

Contact Information - Research staff will collect the following information from participants: (1) contact information; (2) best way to reach an individual if they have more than one line; best times/days to reach participant; and (3) names and contact information of people staff are allowed to contact if participant is lost to follow-up or otherwise cannot be contacted (i.e. collateral contacts). The purpose of this is to maximize the likelihood of reaching a participant to complete the study procedures. Furthermore, asking permission to leave a voicemail on at a specified contact number ensures a greater level of privacy for the participant.

Data Collection - Baseline will take approximately 30 minutes to complete and includes demographic variables, TBI variables (date of injury, TBI severity), medications and information describing participants' pain history, including pain sites, and pain duration. The Brief Pain Intensity measure (BPI), a 4 item pain intensity scale, will be asked 4 times over the course of 7 days at each assessment period.

Follow-up Interviews:

Follow-up interviews will be collected at 4-months and 8-months post-randomization and will each take approximately 45 minutes each.

Collaborative Care

Collaborative Care (CC) is a systematic and integrated approach to improving the delivery and utilization of effective treatments for chronic pain. The care will be delivered through an interdisciplinary team, organized around a CC Manager (CCM) who guides the participant through various aspects of care. The team will include a group of experts on pain and TBI. The CCM will offer all participants care management, collaborative medical management, and psychosocial treatment. If the participant declines to receive any of the components of the intervention, they may still choose to participate in the remaining components.

Usual Care Group

Participants assigned to usual care will be encouraged to consult with their TBI or primary care provider with any concerns around pain treatment. Study personnel will not make any attempts to influence usual care participants' pain management.

Because this is an effectiveness study, treatment decisions for UC participants will be left to the primary provider and may or may not include pharmacologic management, counseling, and referral to specialty services or other local resources.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of mild to severe TBI based on medical chart review;
* Patient has an appointment with the University of Washington/Harborview Medical Center, Department of Rehabilitation Medicine's TBI clinics or has been seen by TBI providers within the last 12 months;
* Patient reports clinically significant pain, defined as having moderate or higher pain over the last 6 months (defined as an average pain score of 4-10/10 on a 0=no pain to 10=worst pain numeric rating scale);
* Patient is "somewhat" or "very" willing to accept additional help with their pain as asked during screening;
* Reads and English speaking (we will track non-enrollment due to other language to determine common languages)
* Has access to and ability to communicate over the phone;
* Aged >18 years of age;
* Provides written informed consent.

Exclusion Criteria:

* Answers more than one incorrect response on the Six-Item Screener;
* Terminal illness or pain associated with cancer diagnosis;
* Major surgery anticipated during study period (approximately 8 months);
* Presence of severe psychiatric disorder as evidenced by high suicide risk, diagnosis of bipolar disorder with psychotic features or current psychotic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from enrollment to end of treament (month 4) in Pain Interference Scale from the Brief Pain Inventory | Collected at 0-14 days of enrollment, Month 4
  A 7-item scale which measures pain interference with general activity, mood, walking, work (outside or in home), relationships, sleep, and enjoyment of life on numerical rating scales (NRS) from 0 (does not interfere) to 10 (interferes completely).

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9)-Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  A measure of depression severity that parallels DSM-5 criteria and has established reliability, validity, and sensitivity to change in people with TBI.
Generalized Anxiety Disorder 7 item (GAD-7) - Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  A measure of general anxiety.
Pittsburgh Sleep Quality Inventory (PSQI) - Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  The PSQI contains 19 items covering 7 dimensions of sleep plus a composite score.
Brief Pain Intensity- 4 (BPI-4) - Change is being assessed. | Collected 4 times in one week over the course of 7 days at enrollment period, Month 4, Month 8
  A 4-item pain intensity scale in past week (current, worst, average, least).
Patient Global Assessment of Treatment Satisfaction (PGATS) - Change is being assessed. | Collected at Month 4, Month 8
  A 3 item measure that rates satisfaction with care received.
Participation Assessment with Recombined Tools - Objective 17 - Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  The PART-O-17 is a patient-reported measure of involvement in life situations at the societal level as reflected in fulfillment of developmentally and culturally appropriate roles such as worker, student, spouse, parent, or citizen.
Cornell Service Index (CSI) - Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  A standardized measure of the quantity and characteristics (for example, site and provider) of health services used.
Visits To Regional Emergency Departments (ED) - Change is being assessed. | Collected at 0-14 days of enrollment, Month 4, Month 8
  Count of visits to regional emergency departments in the last 4 months.
Change from enrollment to 4 months post randomization (month 8) in Pain Interference Scale from the Brief Pain Inventory | Collected at 0-14 days of enrollment, Month 8
  A 7-item scale which measures pain interference with general activity, mood, walking, work (outside or in home), relationships, sleep, and enjoyment of life on numerical rating scales (NRS) from 0 (does not interfere) to 10 (interferes completely).
Chronic Pain Acceptance Questionnaire (CPAQ-8) | Collected at 0-14 days of enrollment, Month 4, Month 8
  An 8-item measure looking at the acceptance of chronic pain
DFAQ-CU Inventory | Collected at 0-14 days of enrollment, Month 4, Month 8
  DFAQ-CU is a 4-item measure and stands for daily sessions, frequency, age of onset, and quantity of cannabis use.
AUDIT-C | Collected at 0-14 days of enrollment, Month 4, Month 8
  A 3-item alcohol screen that can help identify persons who have active alcohol use disorders.
The two-Item Conjoint Screen (TICS) | Collected at 0-14 days of enrollment, Month 4, Month 8
  A two-Item Conjoint Screen, is composed of two questions on alcohol/drug use in the past year and feeling the need to cut down on this use.
Patient Global Impression of Change (PGIC) | Collected at 0-14 days of enrollment, Month 4, Month 8
  A self-report measure which reflects a patient's belief about the efficacy of treatment.
Pain Quality Assessment Scale (PQAS) | Collected at 0-14 days of enrollment, Month 4, Month 8
  Measures different types of pain people may experience.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Hoffman, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, TBI Clinic, Seattle, Washington
  - University of Washington Medical Center, TBI Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curran MC, Lucas S, Fann JR, Zumsteg JM, Hoffman JM. Chronic pain after traumatic brain injury: a collaborative care approach. Front Rehabil Sci. 2024 Aug 26;5:1398856. doi: 10.3389/fresc.2024.1398856. eCollection 2024. PMID 39253025
- [Derived] Hoffman JM, Curran M, Barber J, Lucas S, Fann JR, Zumsteg JM. Collaborative Care for Chronic Pain After Traumatic Brain Injury: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2413459. doi: 10.1001/jamanetworkopen.2024.13459. PMID 38829619